CLINICAL TRIAL: NCT03239990
Title: Group-based Parenting Program "Incredible Years" to Reduce Child Conduct Disorder Symptoms in Families With Child Protection and Other Family Support Services in Finland
Brief Title: Group-based Parenting Program to Reduce Child Conduct Disorder Symptoms in Finland
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Piia Karjalainen, Senior Researcher, Finnish Institute for Health and Welfare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: THL/1059/6.02.01/2015
Record Dates: First submitted 2017-06-15; First posted 2017-08-04 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Conduct Disorders in Children
Keywords: Children's mental health; Conduct disorders; Conduct problems; Externalizing problems; Parental Intervention; Groups based intervention; Finland; Social learning theory; Cognitive-behavioral theory
MeSH Terms: conditions — Conduct Disorder

STUDY DESIGN:
Intervention Model Description: Randomize Controlled Trial with intervention and control groups (TAU)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incredible Years, Parent support (Experimental): Incredible Years, Parent group supported by home visiting includes the Incredible Years Parent Training Program, Preschool Basic version, with 18-20 group meetings. Four home visits are added to the program to support parents in practicing new skills and to provide individual practical consultation.
  Interventions: Behavioral: Incredible Years, Parent group supported by home visiting
- Treatment as usual (No Intervention): The control group will receive treatment as usual

INTERVENTIONS:
Behavioral: Incredible Years, Parent group supported by home visiting — Parents are taught to use positive and consistent strategies in reducing child misbehavior
  Arms: Incredible Years, Parent support

SUMMARY:
According to studies, approximately 20% of children having contact with child protection services have conduct disorder. Negative parenting can make this problem even worse. Research has shown Incredible Years Program to be one of the most effective programs to prevent and reduce child conduct problems. This study is an randomized controlled trial, which evaluates the suitability and effectiveness of group-based Incredible Years program in child protection and family support services. The aim of this study is to find out whether this intervention reduces children's psychiatric symptoms, especially conduct symptoms, increases positive parenting and positive interaction between parents and children, and reduces children's and parent's stress and increase well-being. The study will be carried out in 2015-2018. Overall 101 children and 120 parents participate in the study.

DETAILED DESCRIPTION:
1. Introduction Parenting skills and home environment play a major role in children's development and safety, especially in early childhood. Studies have shown that maltreating parents have poor child management techniques, high levels of hostile feelings, reduced emotional responsiveness and escalated verbal aggression. It is apparent that large number of parents receiving child protection services are engaged in parental behaviors that do not decrease child's problems, but instead may be harmful to their children. Since over 80 000 of the children receiving support from child protection services in Finland remain in their homes, the need of effective methods to support parenting is evident.

   Several randomized trials have shown that parent management training programs, which are based primarily on social learning theory, cognitive-behavioral theory, and attachment theory, effectively improve parenting skills, parents' mental health and child conduct problems. These programs build on social learning theory according to which parents model the appropriate behavior to their children. Behavioristic principles, however, include methods of prompting children's positive behavior. Ideas based on cognitive theory help parents change their conceptions of the child and his/her problematic behavior and coaches them to use problem solving and anger management skills. The basis of attachment theory is that when a sensitive and safe attachment has developed between the child and the caretaker, it helps a child feel safe and builds his/her positive perception of different situations.

   Incredible Years Parent Training Program(IY) is one of the most researched programs and has been found to be effective in different countries and contexts, for example among high-risk, disadvantaged, and maltreating families and also among foster carers . However, only a few studies have been made in the context of child protection services or with maltreated children.

   The IY program is group-based, focuses on building support networks and decreasing isolation, and has a format designed to reduce stigma, and increase parental participation and engagement. It emphasizes individual goal-setting and a self-reflective learning style, as well as intensive behavior practice and rehearsal methods with other parents and a positive, collaborative relationship between group leaders and parents. For the previous reasons it may be particularly relevant to families with child protection services contact and should be thoroughly researched.
2. Aims

   The main study question is:

   Does the group based, intensive Incredible Years Parent Management Training reduce children's (age 3-7) (sub)clinically significant behavioral problems?

   The other study questions are:

   Does Incredible Years Parent Management Training
   * increase positive parenting?
   * increase positive interaction between parents and children?
   * reduce children's (age 3-7) other psychiatric symptoms?
   * reduce children's and parent's stress?
   * increase parent's well-being?
3. Study Design Randomized controlled trial design will be used (RCT). Participants are 3-7 year old children (index children, n=101) with behavioral problems and their parents who are currently clients of child protection services, other special support services for families or families who are clients of family centers or need support just for their parenting. Parents and children were randomized before the baseline measurements to the intervention group or treatment as usual / waiting list condition. The intervention program is Incredible Years Parent Training (Preschool Basic), with 20 parent group meetings, including 4 home visits. Children themselves do not participate in any intervention. Based on earlier studies the intervention effects of parent management training is mediated by changed parenting practices towards children. The measuring points are pre, post and 1 year. The study will be carried out in 2015-2018.

   Intervention Participants will attend the Incredible Years Parent Training Program, Preschool Basic version, with 18-20 group meetings. The program is based mainly on cognitive-behavioral and social learning theories.

   The goal of the group is to enhance and support parenting skills, increase knowledge of child development, improve child's positive behavior and parent-child interaction. Parents are taught to use more positive and consistent strategies in reducing child misbehavior by watching dvd's, rehearsing and group discussions. Groups consist of 10-12 parents and they get together weekly for app. 2-2,5 hours at a time. Four home visits are added to the program to support parents in practicing new skills and to provide individual practical consultation. Also weekly phone calls are being made to the parents, as part of normal procedure of the program.

   Parents will be interviewed before starting the intervention to explain it fully.

   The intervention groups will start in fall 2016 or beginning of 2017. In each group there will be three trained group leaders, of which two are from family counselling services and one a family worker from child protection services, who also conducts family visits.

   Program fidelity The group leaders will receive supervision from certified peer coach every three weeks and once from a mentor during the duration of the groups. Group leaders will fill out check lists and self-evaluations after every group meeting. Also evaluations from parents after every group meeting will be gathered.
4. Ethics

Parents and children are participating voluntarily in the research. Participants of the intervention group are given concrete information and training about positive parenting methods in a supportive and positive peer group by trained leaders. The participants of the control group can access all the other services and support they are entitled to, other than the intervention program being researched. The restrain and discomfort caused to participants can be considered minor.

Families participating the study have been interviewed and their willingness to participate have been asked beforehand. The group leaders of the intervention will interview the participants of the intervention group and tell about the intervention. The participants of the control group have a possibility access the next available parent group in the community.

Parents participating the research have at any time a right to withdraw from the research. Confidentiality will be taken care of.

ELIGIBILITY:
Inclusion Criteria:

* Parents of the child are evaluated by child protection services to benefit from parenting support, or who receive special support for parenting
* Child is between the ages 3-7 when entering the program
* The child is living at home
* Child has behavioral problems
* Parents have the motivation to attend the groups
* There is no unresolved acute child protection issue (child's basic needs and safety are not fulfilled).

Exclusion Criteria:

* Parents have a mental health or substance abuse problem that prevents attending the group.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change in ECBI (Eyberg Child Behavior Checklist) | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 0-3 months after the intervention is finished.
  Change of problem behavior measured by ECBI
Change in CBCL (Child Behaviour Checklist) Externalizing scale | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 0-3 months after the intervention is finished.
  Change of problem behavior measured by CBCL Externalizing scale
Long term change in ECBI | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 12-15 months after the intervention is finished.
  Long term change of problem behavior measured by ECBI
Long term change in CBCL Externalizing scale | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 12-15 months after the intervention is finished.
  Long term change of problem behavior measured by CBCL, Externalizing scale

SECONDARY OUTCOMES:
Change in measure of executive functions (measured by KESKY questionnaire) | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 0-3 months after the intervention is finished.
  Change of a child's executive functions (including, attention, impulsivity and motor restlessness measured by KESKY questionnaire)
Change in CBCL total scores | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 0-3 months after the intervention is finished.
  Change in a child's psychiatric problems measured by CBCL total scores
Change in Dyadic Parent-Child Interaction measured by Dyadic Parent-Child Interaction Coding System | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 0-3 months after the intervention is finished.
  Parent-child interaction quality evaluated by coding 10 minutes videos of child-led play and parent-led play
Change in PPI, Parenting Practices Interview | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 0-3 months after the intervention is finished.
  Parent's self evaluation of his/her parenting practices
Change in PSI-4-SF, Parenting Stress Inventory, short version | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 0-3 months after the intervention is finished.
  Parent's self evaluation of his/her parenting related stress
Change in the Marshmallow test | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 0-3 months after the intervention is finished.
  Child's patience to resist temptation to eat a marshmallow candy
Change in child's risk taking behavior in a gambling task | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 0-3 months after the intervention is finished .
  Child's tendency to take risks in a gambling task to win candies
Change in child's trust to another child | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 0-3 months after the intervention is finished.
  Trust Game (Surprise Bag Task) to evaluate does a child trust she/he gets something back if she/he gives a surprise bag to an other child.
Change in Dictator game for children | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 0-3 months after the intervention is finished.
  Altruism, how much the child is willing to give stickers to another child, who doesn't have any.
Long term change in measure of executive functions (measured by KESKY questionnaire) | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 12-15 months after the intervention is finished.
  Change of a child's executive functions (including attention, impulsivity and motor restlessness measured by KESKY questionnaire)
Long term change in CBCL total scores | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 12-15 months after the intervention is finished.
  Change in a child's psychiatric problems measured by CBCL total scores
Long term change in Dyadic Parent-Child Interaction measured by Dyadic Parent-Child Interaction Coding System | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 12-15 months after the intervention is finished.
  Parent-child interaction quality evaluated by coding 10 minutes videos of child-led play and parent-led play
Long term change in PPI, Parenting Practices Interview | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 12-15 months after the intervention is finished.
  Parent's self evaluation of his/her parenting practices
Long term change in PSI-4-SF, Parenting Stress Inventory, short version | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 12-15 months after the intervention is finished.
  Parent's self evaluation of his/her parenting related stress
Long term change in the Marshmallow test | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 12-15 months after the intervention is finished.
  Child's patience to resist temptation to eat a marshmallow candy
Long term change in child's risk taking behavior in a gambling task | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 12-15 months after the intervention is finished.
  Child's tendency to take risks in a gambling task to win candies
Long term change in child's trust to another child | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 12-15 months after the intervention is finished.
  Trust Game (Surprise Bag Task) to evaluate does a child trust she/he gets something back if she/he gives a surprise bag to an other child.
Long term change in Dictator game for children | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 12-15 months after the intervention is finished.
  Altruism, how much the child is willing to give stickers to another child, who doesn't have any.

OTHER OUTCOMES:
Change in GHQ, General Health Questionnaire, for parent | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 0-3 months after the intervention is finished.
  Parent's general psycho-social health
Change in SWEMWBS (Short version of Warwick-Edinburgh Mental Well-being Scale), Positive mental health questionnaire | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 0-3 months after the intervention is finished.
  Parent's self evaluation of his/her mental well being
Change in Heart rate during rest | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 0-3 months after the intervention is finished.
  Both the parent and the child, to evaluate stress, measured during 10 minutes rest
Long term change in GHQ, General Health Questionnaire, for parent | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 12-15 months after the intervention is finished.
  Parent's general psycho-social health
Long term change in SWEMWBS, Positive mental health questionnaire | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 12-15 months after the intervention is finished.
  Parent's self evaluation of his/her mental well being
Long term change in Heart rate during rest | Baseline measure is conducted 0-4 months before starting the intervention and postintervention measure is measured 12-15 months after the intervention is finished.
  Both the parent and the child, to evaluate stress, measured during 10 minutes rest

CONTACTS AND LOCATIONS:
Overall Officials: Piia Karjalainen, M.ED, Study Director — Finnish Institute for Health and Welfare

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karjalainen P, Santalahti P, Aronen ET, Kiviruusu O. Parent- and teacher-reported long-term effects of parent training on child conduct problems in families with child protection and other support services: a randomized controlled trial. Child Adolesc Psychiatry Ment Health. 2021 Feb 11;15(1):7. doi: 10.1186/s13034-021-00358-6. PMID 33573694